CLINICAL TRIAL: NCT06837649
Title: The Effect of Mindfulness-Based Tai Chi Chuan on Mobile Phone Addiction Among Male College Students is Associated With Executive Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital University of Physical Education and Sports, China (Other)
Responsible Party: Principal Investigator, Bai Shuang, Doctor, Beijing Sport University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KM202210029001
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Mobile Phone Addiction Behavior
Keywords: Mobile Phone Addiction Behavior; Executive Function; Cognitive Function

STUDY DESIGN:
Intervention Model Description: The study will select male university students. Inclusion criteria include:
  Male students not majoring in physical education. Aged 18 years or older. Moderate mobile phone dependence, with a score above 40 on the Mobile Phone Addiction Index (MPAI).
  No regular exercise habits. Willing to participate in an 8-week mindfulness-based Tai Chi training and sign informed consent.
  No serious medical conditions. The control group will not receive any special exercise intervention, while the experimental group will undergo an 8-week mindfulness-based Tai Chi intervention. Participants' mobile phone addiction, mindfulness levels, and executive functions will be assessed before and after the intervention. The study will explore the potential mechanisms by which mindfulness-based Tai Chi improves mobile phone addiction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The exercise time lasts 40 min each time, including 5 min of wuji pile practice with positive thoughts, 30 min of eight styles of Tai Chi Chuan practice (4 min*6 sets, 1 min interval between sets), and 5 min of relaxation part of wuji pile with music. The exercise frequency is 3 times a week.
  Interventions: Behavioral: The mindfulness-based Tai Chi Chuan
- Control group (No Intervention): The control group maintained their normal physical activity levels without any additional intervention.

INTERVENTIONS:
Behavioral: The mindfulness-based Tai Chi Chuan — Studies have shown that compared with the Tai Chi Chuan, MTCC is more relaxing to practitioner. The Tai Chi Chuan section is based on the Yang's movements, which not only conform to the basic technical characteristics, such as the steps, stance, techniques, movement of the center of gravity, and the coordination of the whole body between the movements, but also are clear, smooth, simple, easy to learn, and beautiful. The mindfulness section is complemented by soothing, soft music to guide the practitioner to focus on himself and return to inner peace. The essence of the program is to help practitioners focus their attention and achieve inner peace during practice. Through the practice of MTCC, practitioners are encouraged to face the difficulties they encounter in reality and to develop a positive and open mind to deal with negative emotions and thoughts in daily life.
  Arms: Experimental group

SUMMARY:
The goal of this clinical trial is to investigate whether an 8-week mindfulness-based Tai Chi intervention can improve cognitive and executive functions, particularly inhibitory control, and reduce mobile phone addiction in male university students. It will also explore the potential mechanisms by which mindfulness-based Tai Chi affects mobile phone addiction behaviors. The main questions it aims to answer are:

Does mindfulness-based Tai Chi improve inhibitory control and reduce mobile phone addiction in male university students? Does mindfulness-based Tai Chi enhance overall executive functions, including inhibition, updating, and shifting abilities? Researchers will compare the experimental group (receiving mindfulness-based Tai Chi intervention) to the control group (maintaining their usual routine without intervention) to see if mindfulness-based Tai Chi leads to greater improvements in cognitive and executive functions and reduces mobile phone addiction.

Participants will:

Practice mindfulness-based Tai Chi for 8 weeks Complete pre- and post-intervention assessments of mobile phone addiction, mindfulness levels, and executive function Engage in weekly Tai Chi practice sessions Complete self-report diaries of mobile phone usage and mindfulness experiences

ELIGIBILITY:
Inclusion Criteria:

* Male university students not majoring in physical education. Aged 18 years or older. A moderate level of dependence on mobile phones, with a score above 40 on the Mobile Phone Addiction Index (MPAI).

No regular exercise habits in daily academic life. Willing to participate in an 8-week mindfulness-based Tai Chi training program and provide informed consent.

No serious medical conditions.

Exclusion Criteria:

* The exclusion criteria include individuals with diseases that may affect training (such as cardiovascular diseases, respiratory diseases, and musculoskeletal disorders), as well as those diagnosed with mental disorders (such as depression, anxiety, obsessive-compulsive disorder, etc.).

Ages: 18 Years to 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 66 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-06-03 (Actual)

PRIMARY OUTCOMES:
Mobile Phone Addiction Index | From enrollment to the end of treatment at 8 weeks.
  Measurement of mobile phone addiction used the Mobile Phone Addiction Index (MPAI) developed by Y.K. Leung, which is suitable for measuring mobile phone addiction in college students with a good reliability of 0.87. There are four dimensions in the scale, namely loss of control, withdrawal, avoidance, and ineffectiveness. It is rated from 1 to 5 with 17 questions.
Mindfulness level | From enrollment to the end of treatment at 8 weeks.
  The Mindful Attention Awareness Scale (MAAS) was used to measure the mindfulness level. It developed by Brown and Ryan in 2003, which was introduced and revised by domestic scholars in 2012. Besides, it has high validity, structure validity and retest reliability of 0.87 0.89. The scale of single dimension scale, score from 1 to 6 points, are all positive ratings, which includes 15 problem. The higher the total score is, the higher levels one's mindful awareness and attention are.
Executive Functions | From enrollment to the end of treatment at 8 weeks.
  Executive function was measured by the executive function test instrument developed by Chen Aiguo, whose reliability has been tested in numerous studies. The test consisted of a Flanker task (inhibition function), a 2-back task (updating function), and a More-odd shifting task (shifting function).

CONTACTS AND LOCATIONS:
Locations (1):
- Capital University Of Physical Education And Sports, School of Kinesiology and Health, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD collected throughout the trial,We are willing to share the following data from the participants in the experiment: mobile phone addiction index, mindfulness level, executive functions, and other related information.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD will be made publicly available 6 months after the publication of the paper. The data will be shared on the China National Center for Bioinformation (https://ngdc.cncb.ac.cn/gsub/) for other researchers to access and use. The shared data will include all experimental data that is not related to personal privacy, adhering to data confidentiality and ethical standards.
Access Criteria: After data collection, the data will be entered into the China National Center (https:/ngdc.cncb.ac.cn/gsub/), which is an internet-based electronic data capture and management system. It is used for storing, organizing, and managing research data to ensure the security, accuracy, and traceability of the data
URL: https://ngdc.cncb.ac.cn/gsub/